CLINICAL TRIAL: NCT05054179
Title: The Efficacy of Pecto-intercostal Fascial Plane Catheters for Reduction of Sternal Pain in Cardiac Surgery Patients With Complete Median Sternotomy: A Randomized, Placebo-controlled Trial
Brief Title: Pecto-Intercostal Fascial Plane Block Catheter Trial for Reduction of Sternal Pain
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ron Ree, Clinical Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PIFB Catheter RCT
Record Dates: First submitted 2021-08-19; First posted 2021-09-23 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Cardiac Surgery; Sternotomy; Acute Pain
Keywords: Pecto-intercostal fascial plane catheters; Cardiac surgery; Heart surgery; Sternotomy; Acute pain; Post-sternotomy pain; Chronic Pain
MeSH Terms: conditions — Acute Pain; Chronic Pain | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: This will be a prospective, randomized, triple-blinded, placebo-controlled trial in which patients will be randomly allocated to two study groups on a 1:1 basis into:
  1) Intervention Group: 20 mL of ropivacaine 0.2% will be bolused through PIFB catheters on each side, followed by 3 mL/hour infusion of ropivacaine 0.2% for 48 hours each side.
  2) Control Group: 20 mL of ropivacaine 0.2% will be bolused through PIFB catheters on each side, followed by 3 mL/hour infusion of normal saline for 48 hours each side.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patient Masking: Patients will be informed that they will receive one of two solutions (ropivacaine or saline) for infusion, without disclosing which group they are allocated to.
  Anesthesiologists, cardiac surgeons, Cardiac Surgery Intensive Care Unit (CSICU) nurses, ward nurses, nurse practitioners, and acute pain service team Masking: blinded/masked to assignments.
  Assessors Masking: Assessment of patients, data collection, and follow-up will be conducted by team members (i.e. research assistant, anesthesiologist, CSICU nurses, and ward nurses, acute pain service team) will be blinded/masked to group allocation of a patient participant.
  Data Analyst Masking: The data analysts will be provided a table with two groups of the unique numbers, but which group corresponds with ropivacaine and which corresponds with normal saline will not be revealed until the data analysis has been fully completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The participants of this group will receive 20 mL of 0.2% Ropivacaine via parasternal multi-orifice catheters on each side of the sternum, followed by infusion of 3 mL/h for 48 hours.
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution Bolus; Drug: Ropivacaine 0.2% Injectable Solution Infusion
- Placebo group (Placebo Comparator): The participants of this group will receive 20 mL of 0.2% Ropivacaine via parasternal multi-orifice catheters on each side of the sternum, followed by infusion of 3 mL/h of normal saline for 48 hours.
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution Bolus; Other: Normal Saline Infusion

INTERVENTIONS:
Drug: Ropivacaine 0.2% Injectable Solution Bolus — 20 mL of ropivacaine 0.2% will be injected via parasternal multi-orifice catheters on each side
Other: Normal Saline Infusion — 3 mL/hour infusion of normal saline for 48 hours via parasternal multi-orifice catheters on each side of the sternum
  Arms: Placebo group
Drug: Ropivacaine 0.2% Injectable Solution Infusion — 3 mL/h infusion of Ropivacaine 0.2% for 48 hours via parasternal multi-orifice catheters on each side of the sternum
  Arms: Intervention Group

SUMMARY:
One of the most painful aspects of open heart surgery is the incision made through the skin and the sternum to access the heart (a "sternotomy"). Post-sternotomy pain is a potentially debilitating complication of surgery that slows recovery immediately after surgery and can lead to issues with chronic pain. Previous research has shown that by injecting local anesthesia in the pecto inter-fascial plane, the space between the pectoralis major and the intercostal muscles, pain relief can be provided. The investigators aim to assess if repeated injections of local anesthesia via catheters is a useful adjunct compared to routine care.

DETAILED DESCRIPTION:
Justification:

Post-sternotomy pain after cardiac surgery can be debilitating, with associated risks of decreased respiratory function and chronic pain. Severe acute sternal pain after cardiac surgery occurs in 49% of patients at rest and 78% of patients during coughing. Post-sternotomy pain is worst during the first two days and improves thereafter.

The sternum is innervated by the medial division of the anterior cutaneous branches of the T2-6 intercostal nerves, which may be targeted by several regional anesthetic techniques. Concerns of rare epidural hematoma and possible case cancellations with a bloody tap, in the context of systemic heparinization for cardiac surgery, deters many from utilizing neuraxial analgesia for post-sternotomy pain. Contrarily, parasternal regional blocks such as pecto-intercostal fascial plane block (PIFB) provide a low-risk alternative that targets the anterior cutaneous branches of intercostal nerves, and PIFB has been shown to be effective in improving acute post-sternotomy pain.

Nevertheless, single-shot PIFB is limited by its short duration of action, whereas sternotomy pain can remain severe for two postoperative days. Hence, continuous local anesthetic infusion via bilateral PIFB catheters for 48 hours may improve patient pain experience and related outcomes over single shot PIFB.

Objective:

This study aims to evaluate whether, in addition to single shot PIFB, continuous local anesthetic infusion (compared with placebo infusion) through bilateral PIFB catheters reduces acute sternal pain at 24 hours after cardiac surgery with complete median sternotomy. The 24-hour time point was chosen as it represents a time where both the post-sternotomy pain is rated as severe, especially with movement and coughing, and the patient is required to start actively participating in the postoperative rehabilitative process.

Hypotheses:

This study hypothesize that, in addition to single shot PIFB, continuous ropivacaine infusion through bilateral PIFB catheters will be more effective than placebo infusion in reducing sternal pain score on standardized coughing at 24 hours after cardiac surgery with complete median sternotomy.

Study Design:

This will be a prospective, randomized, triple-blinded, placebo-controlled trial in which patients will be randomly allocated to two study groups on a 1:1 basis into:

1) Treatment Group: 20 mL of ropivacaine 0.2% will be deposited via parasternal multi-orifice catheters on each side, followed by infusion of 3 mL/h for 48 hours.

2) Control Group: 20 mL of ropivacaine 0.2% will be deposited via parasternal multi-orifice catheters on each side, followed by a saline infusion of 3 mL/h for 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled cardiac surgery patients
* Complete median sternotomy
* Adult (19 years old or older)
* English-speaking

Exclusion Criteria:

1. Preoperative Exclusion Criteria:

   * Patient refusal
   * Emergent surgery
   * Inability to provide consent
   * Expected inability to follow up via telephone
   * Known preoperative coagulopathy

     i) Congenital coagulopathy ii) Congenital platelet disorders iii) Platelet count < 50 x 10^9 iv) International normalized ratio (INR) or activated partial thromboplastin time (aPTT) exceeding the upper range of normal in the absence of anticoagulant use v) Does not include active anticoagulant or antiplatelet use
   * Known predicted post-operative therapeutic anticoagulation within 48 hours.
   * Known skin disease over block insertion site that would prevent catheter securement
   * Known Immunodeficiency including uncontrolled diabetes, as defined by HbA1C of 7.8% or more
   * Known preoperative advanced liver failure (as defined by Child-Pugh B or C)
   * Known preoperative advanced renal failure (as defined by Estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73 m2)
   * Known opioid tolerance (as defined by morphine oral equivalent >60mg for a period of 7 days or longer pre-operatively)
   * Known allergy to local anesthetic, acetaminophen, or hydromorphone
   * Known weight less than 60 kg
   * Any known technical or physical barrier to block catheter placement (i.e., deep brain stimulation pulse generator or other devices, breast or other implants)
2. Postoperative Exclusion Criteria:

   * Postoperative bleeding at time of randomization as defined by:

     i) initial chest tube loss of >350 mL ii) >200 mL per hour loss iii) > 2 mL/kg/hour loss for 2 consecutive hours iv) or requiring return to the operating room for surgical management
   * Hemodynamic instability, as determined by Cardiac Surgery Intensive Care Unit (CSICU) attending anesthesiologist
   * Anticipated mechanical ventilation of more than 24 hours
   * Anesthesiologist unavailable to insert Pecto-Intercostal Fascial Plane Block (PIFB) catheter within 4 hours of CSICU arrival
   * Any known technical or physical barrier to block catheter placement (i.e., deep brain stimulation pulse generator or other devices, breast or other implants)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Post-operative Sternal Pain on coughing at 24 hours. | Post-surgery 24 hours after intervention
  Cardiac Surgery Intensive Care Unit nurses or recovery ward nurses will assess and record Numeric Rating Scale (NRS) sternal pain scores on coughing. Coughing will be elicited with a standardized script for a sitting patient:
  "Please use both hands to hold on to the pillow in front of you to hold your chest in. Take a deep breath in, and give me three coughs in a row"
  The scale is from 0 to 10, with 0 being no pain at all and 10 being the worst pain possible.

SECONDARY OUTCOMES:
Cumulative opioid consumption (in IV morphine equivalents) | Post-surgery at 24 and 48 hours after intervention
  After patient's discharge from hospital, medical record will be reviewed for opioid (in IV morphine equivalents) consumption history.
Post-operative sternal pain severity | Post surgery, every 8 hours after intervention up to 48 hours
  Cardiac Surgery Intensive Care Unit nurses or recovery ward nurses will assess and record Numeric Rating Scale (NRS) sternal pain scores at rest and on coughing up to 48 hours after the intervention.
  Coughing will be elicited with a standardized script for a sitting patient:
  "Please use both hands to hold on to the pillow in front of you to hold your chest in. Take a deep breath in, and give me three coughs in a row".
  The scale is from 0 to 10, with 0 being no pain at all and 10 being the worst pain possible.
  These scores will be recorded every 8 hours.
Nausea or vomiting | Post-surgery within 48 hours of intervention
  After patient's discharge from hospital, medical record will be reviewed for nausea or vomiting and reported as yes or no.
Quality of Recovery-15 score (QoR-15) | Pre-surgery (at enrolment) and Post-surgery at 48 hours
  The research assistant/research coordinator will administer Quality of Recovery-15 score (QoR-15). The QoR-15 includes Part A and Part B. Part A consists of 10 questions regarding how the patient has been feeling in the last 24 hours on a 11-point likert scale from 0 to 10, with 0 being "None of the time" and 10 being "All of the time". Part B consists of 5 questions regarding if the patient has had any of the following in the last 24 hours on the same scale as Part A.
Chronic sternal pain | Post-surgery at 3 months and 6 months
  After patient's discharge from hospital, they will be called at 3 months and 6 months post-surgery and asked about their sternal pain severity on a numeric rating scale of 0-10.
Quality of Life Questionnaire | Pre-operatively (at enrolment), 48 hours after intervention and 3 and 6 months after discharge from hospital
  Participants will complete a quality of life questionnaire, the EQ-5D-5L, preoperatively, at 48 hours, 3 months and 6 months. The first two assessments will be done in person, the 3 and 6 month follow-ups will be done over the phone. The questionnaire consists of 5 dimensions of life (Mobility, Self-Care, Usual Activities, Pain and Discomfort, and Anxiety/Depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Overall Health (EQ-5D VAS) | Pre-operatively (at enrolment), 48 hours after intervention and 3 and 6 months after discharge from hospital
  Participants will report their overall health rating using the EQ-5D Visual Analog Scale (0-100, with 0 being the worst health you can imagine and 100 being the best health you can imagine). This is done preoperatively, at 48 hours, 3 months and 6 months. The first two assessments will be done in person, the 3 and 6 month follow-ups will be done over the phone.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Ree, MD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers.

REFERENCES:
- [Background] Liu V, Mariano ER, Prabhakar C. Pecto-intercostal Fascial Block for Acute Poststernotomy Pain: A Case Report. A A Pract. 2018 Jun 15;10(12):319-322. doi: 10.1213/XAA.0000000000000697. PMID 29293481
- [Background] Lee W, Yan YY, Jensen MP, Shun SC, Lin YK, Tsai TP, Lai YH. Predictors and patterns of chronic pain three months after cardiac surgery in Taiwan. Pain Med. 2010 Dec;11(12):1849-58. doi: 10.1111/j.1526-4637.2010.00976.x. Epub 2010 Oct 28. PMID 21040435
- [Background] van Gulik L, Janssen LI, Ahlers SJ, Bruins P, Driessen AH, van Boven WJ, van Dongen EP, Knibbe CA. Risk factors for chronic thoracic pain after cardiac surgery via sternotomy. Eur J Cardiothorac Surg. 2011 Dec;40(6):1309-13. doi: 10.1016/j.ejcts.2011.03.039. Epub 2011 May 10. PMID 21561786
- [Background] Gust R, Pecher S, Gust A, Hoffmann V, Bohrer H, Martin E. Effect of patient-controlled analgesia on pulmonary complications after coronary artery bypass grafting. Crit Care Med. 1999 Oct;27(10):2218-23. doi: 10.1097/00003246-199910000-00025. PMID 10548210
- [Background] Sasseron AB, Figueiredo LC, Trova K, Cardoso AL, Lima NM, Olmos SC, Petrucci O. Does the pain disturb the respiratory function after open heart surgery? Rev Bras Cir Cardiovasc. 2009 Oct-Dec;24(4):490-6. doi: 10.1590/s0102-76382009000500010. English, Portuguese. PMID 20305922
- [Background] Mueller XM, Tinguely F, Tevaearai HT, Revelly JP, Chiolero R, von Segesser LK. Pain location, distribution, and intensity after cardiac surgery. Chest. 2000 Aug;118(2):391-6. doi: 10.1378/chest.118.2.391. PMID 10936130
- [Background] Lahtinen P, Kokki H, Hynynen M. Pain after cardiac surgery: a prospective cohort study of 1-year incidence and intensity. Anesthesiology. 2006 Oct;105(4):794-800. doi: 10.1097/00000542-200610000-00026. PMID 17006079
- [Background] Milgrom LB, Brooks JA, Qi R, Bunnell K, Wuestfeld S, Beckman D. Pain levels experienced with activities after cardiac surgery. Am J Crit Care. 2004 Mar;13(2):116-25. PMID 15043239
- [Background] Mittnacht AJC, Shariat A, Weiner MM, Malhotra A, Miller MA, Mahajan A, Bhatt HV. Regional Techniques for Cardiac and Cardiac-Related Procedures. J Cardiothorac Vasc Anesth. 2019 Feb;33(2):532-546. doi: 10.1053/j.jvca.2018.09.017. Epub 2018 Sep 13. No abstract available. PMID 30529177
- [Background] Hemmerling TM, Cyr S, Terrasini N. Epidural catheterization in cardiac surgery: the 2012 risk assessment. Ann Card Anaesth. 2013 Jul-Sep;16(3):169-77. doi: 10.4103/0971-9784.114237. PMID 23816670
- [Background] Fujii S, Bairagi R, Roche M, Zhou JR. Transversus Thoracis Muscle Plane Block. Biomed Res Int. 2019 Jul 7;2019:1716365. doi: 10.1155/2019/1716365. eCollection 2019. PMID 31360703
- [Background] Fujii S, Roche M, Jones PM, Vissa D, Bainbridge D, Zhou JR. Transversus thoracis muscle plane block in cardiac surgery: a pilot feasibility study. Reg Anesth Pain Med. 2019 May;44(5):556-560. doi: 10.1136/rapm-2018-100178. Epub 2019 Mar 21. PMID 30902911
- [Background] Chin KJ. An Anatomical Basis for Naming Plane Blocks of the Anteromedial Chest Wall. Reg Anesth Pain Med. 2017 May/Jun;42(3):414-415. doi: 10.1097/AAP.0000000000000575. No abstract available. PMID 28419049
- [Background] Murata H, Hida K, Hara T. Reply to Dr Del Buono et al. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):792. doi: 10.1097/AAP.0000000000000491. No abstract available. PMID 27776104
- [Background] Fujii S, Vissa D, Ganapathy S, Johnson M, Zhou J. Transversus Thoracic Muscle Plane Block on a Cadaver With History of Coronary Artery Bypass Grafting. Reg Anesth Pain Med. 2017 Jul/Aug;42(4):535-537. doi: 10.1097/AAP.0000000000000607. No abstract available. PMID 28632672
- [Background] Garcia Simon D, Fajardo Perez M. Safer alternatives to transversus thoracis muscle plane block. Reg Anesth Pain Med. 2019 Jul 11:rapm-2019-100666. doi: 10.1136/rapm-2019-100666. Online ahead of print. No abstract available. PMID 31300596
- [Background] Fujii S. Transversus thoracis muscle plane block and alternative techniques. Reg Anesth Pain Med. 2019 Jul 11:rapm-2019-100755. doi: 10.1136/rapm-2019-100755. Online ahead of print. No abstract available. PMID 31300594
- [Background] Ueshima H, Otake H. RETRACTED: Optimal site for the subpectoral interfascial plane block. J Clin Anesth. 2017 Feb;37:115. doi: 10.1016/j.jclinane.2016.12.022. Epub 2017 Jan 9. No abstract available. PMID 28235498 (Retraction: PMID 35393192 J Clin Anesth. 2022 Aug;79:110774)
- [Background] McDonald SB, Jacobsohn E, Kopacz DJ, Desphande S, Helman JD, Salinas F, Hall RA. Parasternal block and local anesthetic infiltration with levobupivacaine after cardiac surgery with desflurane: the effect on postoperative pain, pulmonary function, and tracheal extubation times. Anesth Analg. 2005 Jan;100(1):25-32. doi: 10.1213/01.ANE.0000139652.84897.BD. PMID 15616047
- [Background] Gianchandani RY, Saberi S, Zrull CA, Patil PV, Jha L, Kling-Colson SC, Gandia KG, DuBois EC, Plunkett CD, Bodnar TW, Pop-Busui R. Evaluation of hemoglobin A1c criteria to assess preoperative diabetes risk in cardiac surgery patients. Diabetes Technol Ther. 2011 Dec;13(12):1249-54. doi: 10.1089/dia.2011.0074. Epub 2011 Aug 21. PMID 21854260
- [Background] Jokinen MJ, Neuvonen PJ, Lindgren L, Hockerstedt K, Sjovall J, Breuer O, Askemark Y, Ahonen J, Olkkola KT. Pharmacokinetics of ropivacaine in patients with chronic end-stage liver disease. Anesthesiology. 2007 Jan;106(1):43-55. doi: 10.1097/00000542-200701000-00011. PMID 17197844
- [Background] Christensen MC, Dziewior F, Kempel A, von Heymann C. Increased chest tube drainage is independently associated with adverse outcome after cardiac surgery. J Cardiothorac Vasc Anesth. 2012 Feb;26(1):46-51. doi: 10.1053/j.jvca.2011.09.021. Epub 2011 Nov 18. PMID 22100857
- [Background] Bernstein SL, Bijur PE, Gallagher EJ. Relationship between intensity and relief in patients with acute severe pain. Am J Emerg Med. 2006 Mar;24(2):162-6. doi: 10.1016/j.ajem.2005.08.007. PMID 16490644
- [Background] Zubrzycki M, Liebold A, Skrabal C, Reinelt H, Ziegler M, Perdas E, Zubrzycka M. Assessment and pathophysiology of pain in cardiac surgery. J Pain Res. 2018 Aug 24;11:1599-1611. doi: 10.2147/JPR.S162067. eCollection 2018. PMID 30197534
- [Derived] Jen TTH, Prabhakar C, Matras PJ, Rondi K, Bruce S, Sun T, Edwards NY, Mehta S, Schwarz SKW, Chau A, Ree RM. Analgesic efficacy of continuous superficial parasternal intercostal plane blockade in patients undergoing cardiac surgery with median sternotomy: a randomized controlled trial. Reg Anesth Pain Med. 2025 Nov 26:rapm-2025-107162. doi: 10.1136/rapm-2025-107162. Online ahead of print. PMID 41193383
- See also: Opioid Analgesic Risk Evaluation and Mitigation Strategy (REMS) by U.S. Food and Drug Administration — http://www.fda.gov/drugs/information-drug-class/opioid-analgesic-risk-evaluation-and-mitigation-strategy-rems

DOCUMENTS (1):
  • Study Protocol (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/79/NCT05054179/Prot_003.pdf